CLINICAL TRIAL: NCT02585011
Title: Effect of Local Infiltration Anesthesia With Ropivacaine on Postoperative Pain After Hip Hemiarthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015/1201
Record Dates: First submitted 2015-10-14; First posted 2015-10-23 (Estimated); Last update posted 2020-09-11 (Actual); Status verified 2020-09

CONDITIONS: Femoral Neck Fractures
Keywords: Hemiarthroplasty; Anesthesia, Local; Pain, Postoperative
MeSH Terms: conditions — Femoral Neck Fractures; Pain, Postoperative | interventions — Ropivacaine; Epinephrine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Experimental): Local infiltration anesthesia, single shot during surgery. 150 ml Ropivacaine (2mg/ml), added 0.5 ml Epinephrine (1mg/ml)
  Interventions: Drug: Ropivacaine; Drug: Epinephrine
- Placebo (Placebo Comparator): Single shot during surgery.150 ml saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Ropivacaine
  Arms: Ropivacaine
Drug: Epinephrine
  Arms: Ropivacaine
Drug: Saline
  Arms: Placebo

SUMMARY:
At St.Olavs Hospital each year about 400 patients are treated for femoral neck fractures, 250 of them receiving hemiarthroplasty. Implementation of fast-track clinical pathways reduces morbidity and enhances recovery of patients undergoing hemiarthroplasty. One of the key prerequisites for early rehabilitation is optimized pain relief. Local infiltration anesthesia with Ropivacaine is part of a multimodal pain regimen for patients receiving hemiarthroplasty at St.Olavs Hospital, although the pain reducing effect of local Ropivacaine after hemiarthroplasty has not been investigated in clinical trials. In this study it will be investigated whether a single shot with Ropivacaine reduces acute postoperative pain and opioid requirement after hemiarthroplasty. The findings of this study will have a direct impact on patient treatment.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for hemiarthroplasty at St. Olavs Hospital
* competent and willing to give consent
* able to be mobilized in the PACU and in the trauma ward unit.

Exclusion Criteria:

* contraindications for spinal anesthesia, Dexamethasone, Dolcontin or Acetaminophene
* receiving general anesthesia
* patients operated on with an approach different to standard direct lateral surgery
* receiving osteosyntheses
* receiving femoral block less than 4 hours before surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2018-05-13 (Actual); Study Completion 2018-05-13 (Actual)

PRIMARY OUTCOMES:
Pain sensation during mobilization in the post-anesthesia care unit. | 24 hours (day of surgery)
  Pain is registered using the numeric rating scale (NRS) by the nurses both during rest and mobilization. The patients are asked a standard question; on a scale from 0 to 10, where 0 is no pain and 10 is the worst imaginable pain, can you define the pain you have right now?

SECONDARY OUTCOMES:
Pain during mobilization on the day after surgery | 48 hours (first postoperative day)
  Pain is registered using the numeric rating scale (NRS) by the nurses both during rest and mobilization. The patients are asked a standard question; on a scale from 0 to 10, where 0 is no pain and 10 is the worst imaginable pain, can you define the pain you have right now?
Total consumption of opioids on the first postoperative day | 48 hrs (first postoperative day)

CONTACTS AND LOCATIONS:
Overall Officials: Olav Foss, Phd, Study Director — Ortopedisk forskningssenter, St.Olavs Hospital
Locations (1):
- Ortopedisk forskningssenter, St.Olavs Hospital, Trondheim, Norway